CLINICAL TRIAL: NCT03404830
Title: Effects of a Program of High Intensity Exercise by Intervals on the Risk of Falls the Physical Condition and the State of Health in People Over 60 Years
Brief Title: High Intensity Training to Reduce the Risk of Falls in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal Investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Jaén
Record Dates: First submitted 2017-12-05; First posted 2018-01-19 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-01

CONDITIONS: Risk of Falls

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Groups were assigned during the months of July and August through the sports centers where these elderly people performed some kind of physical activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT group (Experimental): This group receives physical training based on HIIT
  Interventions: Other: HIIT group, MICT group
- MICT group (Experimental): This group receives physical training based on MICT
  Interventions: Other: HIIT group, MICT group
- No intervention group (No Intervention): This group does not receive any treatment.

INTERVENTIONS:
Other: HIIT group, MICT group — The HIIT program training:
  5 minutes of heating will be done. The intervention will consist of a training in suspension (TRX) performing squats. The session will be divided into four four-minute intervals at an intensity of 90-95% of the maximum heart rate, followed by three-minute active rest intervals of 50-70%. This intensity will be assigned to each subject individually. After the training, there will be a return to calm of 10 minutes of exercises of joint range. There will be 2 weekly training, with three days between both training, for a period of 12 weeks.
  The training of the MICT program:
  5 minutes of heating will be done. Subsequently, participants will perform a squat training with the Suspension Training System (TRX) with an intensity close to 70% of their maximum heart rate maintained for 40 minutes. The session will conclude with a return to calm of 10 min of joint width and stretching.
  Arms: HIIT group; MICT group

SUMMARY:
Due to the high incidence of falls in the elderly population, this study is presented as a method to reduce the risk of falls through a specific type of training in people over 60 years of age.

DETAILED DESCRIPTION:
A 16-week high intensity interval training (HIIT) program, compared to a continuous exercise program and one that does not perform any training program, decreases the risk of falls and improves the state of health, physical condition and quality of life to a greater extent than a group that does not perform any type of exercise in people over 60 years.

ELIGIBILITY:
Inclusion Criteria:

* To participate in the study, participants will be required to be 60 years of age or older.

Exclusion Criteria:

* All participants with diseases that may alter balance and functional activity (such as auditory or vestibular alterations), central or peripheral neurological disorders, other rheumatological diseases, or serious psychiatric or somatic diseases will be excluded.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Opto-electric measuring system. | Up to twelve weeks.
  To be used to control the parameters of the gait.
CT10P | Up to twelve weeks.
  Can be used for the assessment of dynamic equilibrium, which aims to walk ten steps followed by a straight line on the ground, in the shortest time possible, without losing speed, or support a cake off the line.
UPDATE AND PERFORM THE TEST | Up to twelve weeks.
  Be employed for the assessment of dynamic balance, in which the subject starts from the sitting position in a chair (without palm rest). The evaluator's verbal signal initiates time control (sec). The evaluator must: get up from the chair, travel a distance of 3 meters, go around a pivot, travel the same distance back and sit back in the chair as quickly as possible. The closing of the time is established when the evaluated subject makes contact with the chair sitting down.
Sensor Medica | Up to twelve weeks.
  It has been used to measure the static equilibrium and the calculation of the displacement of the center of pressures (CoP).
Opto-electric measurement system | Up to twelve weeks.
  It has been used for the evaluation of the reaction speed of the lower train and the upper train of the participants, with three different tests, acoustic, optical and optoacoustic.
Dynamometer | Up to twelve weeks.
  Be used to assess the muscle strength of each participant in your dominant hand.
Confidence Scale of the specific balance of activities (ABC) | Up to twelve weeks.
  Be used to assess the fear of falling.
Falls Efficacy Scale-International (FES-I) | Up to twelve weeks.
  Be used to assess the confidence in carrying out daily activities of the participants.
Pulsometer | Up to twelve weeks.
  It will be used to measure the heart rate of the participants in the performance of a cardiorespiratory function test.
UKK walk test of 2 km | Up to twelve weeks.
  It will be necessary to assess the cardiorespiratory frequency of the participants in a walking test 2 km as fast as possible.
InBody 720 | Up to twelve weeks.
  It will be used for the assessment of the lean muscle mass, the segmental fat mass and the amount of intra and extracellular water.
SF-36 (The Short Form-36 Health Survey) | Up to twelve weeks.
  Will be used to assess the quality of life in its Spanish version.
HADS (Hospital Anxiety And Depression Scale) | Up to twelve weeks.
  It will be used to evaluate the depression and anxiety levels of the participants.
Accelerometer | Up to twelve weeks.
  It will be used to assess the quality of sleep, control of the period of physical activity, sedentary period and energy expenditure.

CONTACTS AND LOCATIONS:
Locations (1):
- AQUASPORT PIZARRA pool, Pizarra, Málaga, Spain

REFERENCES:
- [Derived] Jimenez-Garcia JD, Hita-Contreras F, de la Torre-Cruz MJ, Aibar-Almazan A, Achalandabaso-Ochoa A, Fabrega-Cuadros R, Martinez-Amat A. Effects of HIIT and MIIT Suspension Training Programs on Sleep Quality and Fatigue in Older Adults: Randomized Controlled Clinical Trial. Int J Environ Res Public Health. 2021 Jan 29;18(3):1211. doi: 10.3390/ijerph18031211. PMID 33572909